CLINICAL TRIAL: NCT01113996
Title: Optimization of Monitoring Patients Who Are Obese Surgery for Gastric By-pass Protein Supplementation and Physical Training: Interventional Randomized Trial
Brief Title: Monitoring Patients Who Are Obese Surgery for Gastric By-pass Protein Supplementation and Physical Training (PROMISE)
Acronym: PROMISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P081108
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: Obesity; Gastric by-pass; Body composition; Nutrition; Physical activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard treatment - usual care (No Intervention)
- Protein supplementation (Experimental)
  Interventions: Dietary Supplement: Protein supplementation
- Protein supplementation and strength training (Experimental)
  Interventions: Behavioral: Protein supplementation and strength training

INTERVENTIONS:
Behavioral: Protein supplementation and strength training — Protein supplementation and strength training
  Arms: Protein supplementation and strength training
Dietary Supplement: Protein supplementation — Protein supplementation
  Arms: Protein supplementation

SUMMARY:
The purpose of the study is to test whether additional protein intake with or without strength training will help to maintain body composition (fat-free mass) after surgical treatment of obesity by gastric by pass. The main hypothesis is that additional protein intake will limit fat-free mass loss during surgery-induced weight loss, and that strength training will have an additional beneficial effect

DETAILED DESCRIPTION:
Design: Open randomised controlled trial comparing, in obese patients after GBP, an additional oral intake of protein with or without a muscular-strengthening physical training programme (18 weeks) to standard medical and nutritional follow-up after bariatric surgery as control (3 groups). Primary outcome: Variation at 6 months after GBP in total and appendicular fat-free mass as assessed by dual-energy X-ray absorptiometry (DXA). Duration of the study: 36 months. Duration of participation for one patient: 7 months. Number of centers: Monocentric study.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age between 18 and 60 years
* Planned obesity treatment by gastric bypass
* Written informed consent

Exclusion Criteria:

* Subject not affiliated with a social security scheme
* Refusal
* Regular follow-up not feasible
* Participation in a structured physical activity program
* Recent coronary event
* Uncontrolled hypertension
* proliferative diabetic retinopathy or disabling neuropathy, treatment by dialysis, orthopedic problems
* Pregnancy
* Specific food intolerance to protein products
* Abnormal cardiac stress test

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2010-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in fat-free mass at 6 months | 6 months

SECONDARY OUTCOMES:
Variation at 6 months after GBP of other body composition components | 6 months
Variation at 6 months after GBP in dietary habits | 6 months
Variation at 6 months after GBP in muscular strength and habitual physical activity | 6 months
Variation at 6 months after GBP in quality of life and obesity co-morbidities | 6 months
Variation at 6 months after GBP in obesity-associated inflammatory markers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel OPPERT, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- GH-Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Bellicha A, Ciangura C, Roda C, Torcivia A, Portero P, Oppert JM. Changes in Cardiorespiratory Fitness After Gastric Bypass: Relations with Accelerometry-Assessed Physical Activity. Obes Surg. 2019 Sep;29(9):2936-2941. doi: 10.1007/s11695-019-03932-2. PMID 31073952
- [Derived] Oppert JM, Bellicha A, Roda C, Bouillot JL, Torcivia A, Clement K, Poitou C, Ciangura C. Resistance Training and Protein Supplementation Increase Strength After Bariatric Surgery: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 Nov;26(11):1709-1720. doi: 10.1002/oby.22317. PMID 30358153